CLINICAL TRIAL: NCT00894647
Title: A Phase 3b Randomized, Double-blinded, Placebo-controlled, Multicenter, Efficacy and Safety Study of Imiquimod Cream Following Cryosurgery for the Treatment of Actinic Keratoses
Brief Title: Safety and Effectiveness Study of Actinic Keratosis Treatment Following Cryosurgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Sharon Levy, MD, Graceway Pharmaceuticals, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW01-0901
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2010-08-23 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; skin disease
MeSH Terms: conditions — Keratosis, Actinic; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): placebo cream in 250mg/packet, up to 2 packets applied daily
  Interventions: Drug: placebo cream
- imiquimod cream (Active Comparator): Imiquimod 3.75% cream, 250 mg single-use packets, up to 2 packets applied daily
  Interventions: Drug: imiquimod cream

INTERVENTIONS:
Drug: imiquimod cream — Imiquimod 3.75% cream (250 mg/packet) up to 2 packets applied daily Two 2-week treatment periods (Cycle 1 and Cycle 2) separated by a 2-week no-treatment period
  Arms: imiquimod cream
Drug: placebo cream — cream applied once daily for two 2-week treatment periods (Cycle 1 and Cycle 2) separated by a 2-week no-treatment period
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of imiquimod cream versus placebo cream when used after cryosurgery in the treatment of actinic keratoses (AKs).

DETAILED DESCRIPTION:
In this multicenter, randomized, double-blind, placebo-controlled study, the efficacy and safety of imiquimod 3.75% cream following cryosurgery to treat clinically typical visible or palpable AK lesions on the face was compared with that of placebo cream. Based on a 1:1 randomization, approximately 120 subjects applied imiquimod 3.75% cream daily (up to 500 mg cream daily [18.75 mg imiquimod]) and approximately 120 subjects applied placebo cream daily during two 2-week periods (Cycle 1 and Cycle 2) separated by 2 weeks of no treatment. Subjects visited the clinic 9 times-1 screening/cryosurgery visit (additional visits might be needed during the screening period to assess healing from the cryosurgery), 4 treatment visits(treatment initiation at Weeks 0 and 4 and treatment follow-up at the end of Weeks 2 and 6), and 4 posttreatment visits (4, 8, 14, and 20 weeks after the last administration of study treatment at the end of Week 6). The total study duration for a subject, including a 2-week screening period, was up to 28 weeks.

Prior to cryosurgery, subjects had to have ≥10 clinically typical visible or palpable AK lesions in an area that exceeded 25 cm^2 on the face to be eligible for participation in the study. At screening, a minimum of 5 visible lesions were not treated with cryosurgery, and 5 to 14 visible lesions were treated with cryosurgery. Subjects had to have at least 5 AK lesions after the skin healed sufficiently from the cryosurgery to be eligible for randomization to either imiquimod 3.75% or placebo cream. Subjects applied up to 2 packets of study cream (500 mg total) as a thin layer to the entire face, avoiding the periocular areas, lips, and nares; ears were excluded from both assessment and treatment. Study cream was applied prior to normal sleeping hours and removed approximately 8 hours later with mild soap and water. Rest periods from daily treatment could be approved by the investigator as needed, with treatment resumption at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Negative urine pregnancy test (for women of child-bearing potential) and agree to use an approved method of birth control while enrolled in the study.
* Prior to cryosurgery, have ≥ 10 clinically typical (visible or palpable) AKs in an area that exceeds 25 cm2 on the face.
* Must have had cryosurgery on 5 to 14 AKs on the face after giving informed consent and prior to receiving study medication. Lesions previously treated with cryosurgery must be healed sufficiently prior to randomization to study cream.
* Following cryosurgery, have ≥ 5 clinically typical (visible or palpable) AKs in an area that exceeds 25 cm2 on the face that are suitable for treatment with the study cream.

Exclusion Criteria:

* Women who are pregnant, lactating, or planning to become pregnant during the study
* Had a medical event within 90 days of the visit (e.g., stroke, heart attack, etc.).
* Have any skin condition in the treatment area that may be made worse by treatment with imiquimod (e.g., rosacea, psoriasis, atopic dermatitis, eczema).
* Have received specific treatments/medications in the treatment area within the designated time period prior to study treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, Study Director — Graceway Pharmaceuticals, LLC
Locations (18):
- United States (14):
  - Dermatology Research Associates, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - Spencer Dermatology & Skin Surgery Center, Saint Petersberg, Florida
  - Palm Beach Dermatology, West Palm Beach, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Evanston Northwestern Healthcare, Skokie, Illinois
  - Skin Specialists PC, Omaha, Nebraska
  - Academic Dermatology Association, Albuquerque, New Mexico
  - DermResearchCenter of New York, Stony Brook, New York
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - DermResearch Inc., Austin, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Canada (4):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Clinique de Dermatologie, Moncton, New Brunswick
  - Ultranova Skincare, Barrie, Ontario
  - Probity Medical Research, Waterloo, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened in 20 sites-16 in the United States of America (U.S.A.) and 4 in Canada. Screening began on 01 Jun 2009 and the last subject was enrolled on 03 Aug 2009.
Pre-assignment Details: Subjects had to have ≥10 AK lesions in an area the face to participate in the study. At screening, at least 5 visible lesions were not treated with cryosurgery, and 5 to 14 visible lesions were treated with cryosurgery. Subjects needed at least 5 AK lesions after the skin healed sufficiently from the cryosurgery to be eligible for randomization.
Groups:
- Placebo Cream: placebo cream in 250 mg/packet, up to 2 packets applied daily
Period: Overall Study
Arm/Group | Placebo Cream | Imiquimod Cream
Started | 121 | 126
Completed | 111 | 112
Not Completed | 10 | 14
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Non-compliance with study procedures | 0 | 2
Not completed — Other, not due to AE | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Cream | Imiquimod Cream | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 63 | 111
  >=65 years | 73 | 63 | 136
Age Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.05) | 66.0 (9.49) | 66.7 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 106 | 108 | 214
Region of Enrollment [Number; unit: participants]
  United States | 90 | 91 | 181
  Canada | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Lesion Count
Description: The primary efficacy endpoint was a comparison between the active and placebo treatment groups of percent change from baseline in the total AK lesion count at Week 26. All AK lesions on the face were included in the analysis-treated and untreated AK lesions at baseline (defined as the AK lesion count just prior to cryosurgery) and new lesions that appeared post-baseline.
Time Frame: Week 26
Population: Intent to treat population, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: percentage of lesion count
Arm/Group | Placebo Cream | Imiquimod Cream
Number analyzed (Participants) | 121 | 126
percentage of lesion count | -43.3 (30.66) | -77.4 (27.54)

2. Secondary Outcome: Percent of Subjects With Complete Clearance
Description: Proportion of subjects who achieved complete clearance of all AK lesions, cryosurgery-treated AK lesions, and non cryosurgery-treated AK lesions from baseline to Week 26/EOS in the ITT population.
Time Frame: Week 26
Population: Intent to treat (ITT) population, last observation carried forward (LOCF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Cream | Imiquimod Cream
Number analyzed (Participants) | 121 | 126
percentage of participants | 3 [0.9 to 8.2] | 30 [22.3 to 39.0]

3. Secondary Outcome: Number of Participants With Any Post-baseline Local Skin Reactions (LSRs)
Description: LSRs were assessed independently from AEs. The frequency and percentage of subjects, as well as the mean (SD) and median score for severity (none=0, mild=1, moderate=2, and severe=3), were summarized by treatment group and by visit for the following LSRs: erythema, edema, weeping/exudates, flaking/ scaling/dryness, and scabbing/crusting. Erosion and ulceration were also evaluated (none=0, erosion=1, and ulceration=2). A score of greater than 0 for the specified LSR was considered a "treatment site reaction".
Time Frame: Weeks 2, 4, 6, 10, 14, 20, and 26
Population: Safety population: all randomized subjects were presumed to have applied at least one application of study medication and were included in the safety population. This population was used for all safety analyses. Subjects were analyzed as treated.
Measure: Number; unit: participants
Arm/Group | Placebo Cream | Imiquimod Cream
Number analyzed (Participants) | 121 | 126
participants
  Edema | 9 | 93
  Erythema | 88 | 125
  Weeping/Exudate | 9 | 64
  Flaking/Scaling/Dryness | 3 | 114
  Scabbing, crusting | 81 | 112
  Erosion/Ulceration | 22 | 60

ADVERSE EVENTS:
Time Frame: Up to the end of study visit - Week 26
Description: AEs were collected from Visit 1 to the end of the final study visit for each subject.
Arm/Group | Placebo Cream | Imiquimod Cream
Serious Adverse Events (participants affected / at risk) | 2/121 | 6/126
Other Adverse Events (participants affected / at risk) | 28/121 | 54/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cream (N=121) | Imiquimod Cream (N=126)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Fractured Leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Worsening of sciatic nerve (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep right thigh bruise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Possible viral syndrome (Infections and infestations) | 0 (0) | 1 (1)
Squamous cell carcinoma right cheek (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (Possible cardiac arrest) (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cream (N=121) | Imiquimod Cream (N=126)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (6)
Application site irritation (General disorders) | 1 (1) | 7 (7)
Application site pain (General disorders) | 0 (0) | 6 (6)
Application site pruritus (General disorders) | 1 (1) | 12 (12)
Fatigue (General disorders) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 7 (7)
Bronchitis (Infections and infestations) | 5 (5) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)

LIMITATIONS AND CAVEATS:
A treatment-emergent AE (TEAE) was an AE that began or worsened in severity after the first application of study drug. TEAEs were summarized for each treatment group by overall incidence, descending order, relationship to study drug, and severity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No